CLINICAL TRIAL: NCT02249598
Title: Competitive Carriage of Neisseria Spp.; Discovering New Methods of Inhibiting Carriage of Neisseria Meningitidis (Lactamica 2)
Brief Title: Competitive Carriage of Neisseria Spp(Lactamica 2)
Acronym: Lactamica 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH16097
Record Dates: First submitted 2014-08-12; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Neisseria Lactamica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Univeristy of Sheffield (Experimental): lactamica
  Interventions: Biological: lactamica
- Hallam University (Placebo Comparator): Phosphate Buffered Saline (PBS)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: lactamica
  Arms: Univeristy of Sheffield
Biological: Placebo
  Arms: Hallam University

SUMMARY:
In the future it is likely that we will replace the current schedule of injected vaccines with interventions that interrupt transmission of infections in more subtle ways. The agent that causes meningococcal disease (Neisseria meningitidis) colonises the nasopharynx of individuals. In most people, the bacterium is harmless and survives for months in the nasopharynx, however in a minority of people the bacteria can cause invasive disease.

Simply reducing colonisation amongst target groups may protect them, and the rest of the population as well. In a previous study we investigated cross protective antibodies, and found incidentally that inoculating adult volunteers with Neisseria lactamica, a harmless 'cousin' of N. meningitidis, possibly prevents N. meningitidis carriage. If true this could lead to novel mechanisms of reducing colonisation in targeted groups, possibly in the form of a nasal medication. The proposed study large experimental challenge study funded by Meningitis UK that will aim to establish if N. lactamica does or does not inhibit colonisation by N. meningitidis. We will also determine whether N. lactamica displaces existing N. meningitidis carriage, and whether there are individuals who are innately resistant to any Neisseria carriage. The study will recruit 300 volunteers between the ages of 1830yrs from the two universities in Sheffield. It will involve placing droplets of N.lactamica bacteria into the nose of half our group of volunteers, and a harmless water like solution into the nose of the other half of volunteers. We will carry out nose swabs at intervals over a six month period to establish if the pattern of N.meningitidis carriage is effected by N.lactamica colonisation. If the findings are positive we will perform future mechanistic investigations. A62.

ELIGIBILITY:
Inclusion Criteria:

* Currently healthy
* Students and university employees from either Sheffield Hallam University or the University of Sheffield between the ages of 18 and 25yrs.
* Fully conversant in the English language
* Able to attend the full protocol timetable

Exclusion Criteria:

* Individuals who are Immunocompromised due to a medical condition
* Individuals taking immune modifying medications (not including inhaled steroids)
* Individuals in close contact with immunocompromised people including medical students with full time clinical attachments.
* Individuals who have an current infection
* Current Smokers
* People with an allergy to yeast extract.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The number of participants found to have carriage of the bacterium Neisseria meningitidis at 6 sampling points (culture of throat swaps) following innoculation as baseline of subjects with the bacterium Neisseria lactamica | number of positive results presenting between day 0 (baseline) until study completion (28 weeks)
  culture of throat swabs at 2 weeks, 4 weeks, 8 weeks, 16 weeks, 26 weeks and 28 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Read, Principal Investigator — Sheffield NHS Trust
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, South Yorskshire, United Kingdom

REFERENCES:
- [Derived] Deasy AM, Guccione E, Dale AP, Andrews N, Evans CM, Bennett JS, Bratcher HB, Maiden MC, Gorringe AR, Read RC. Nasal Inoculation of the Commensal Neisseria lactamica Inhibits Carriage of Neisseria meningitidis by Young Adults: A Controlled Human Infection Study. Clin Infect Dis. 2015 May 15;60(10):1512-20. doi: 10.1093/cid/civ098. Epub 2015 Mar 25. PMID 25814628